CLINICAL TRIAL: NCT06631924
Title: Intramedullary Fixation for Metacarpal Fractures: A Prospective Study Comparing Outcomes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0802
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Metacarpal Fracture
Keywords: fractures metacrapal
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- • Operative Cohort: Patients who undergo hand surgery at University of Colorado Hospital and Denver: • Operative Cohort: Patients who undergo hand surgery at University of Colorado Hospital and Denver Health Medical Center for surgical treatment of closed extraarticular metacarpal fracture(s). Fracture classification will be based off of AO Foundation/Orthopaedic Trauma Association guidelines and radiographic interpretation
  Interventions: Device: Implant

INTERVENTIONS:
Device: Implant — Intramedullary headless hardware systems were utilized to place hardware in85 a retrograde manner from the metacarpophalangeal joint.

SUMMARY:
To prove that use of intramedullary cannulated headless hardware fixation of metacarpal fractures provides anatomic reduction, stable fixation, less operative trauma and early, active post-operative mobilization. The study compares two types of implant to determine efficacy in reduction and maintenance of reduction for fracture healing.

DETAILED DESCRIPTION:
To prove that use of intramedullary cannulated headless hardware fixation of metacarpal fractures provides anatomic reduction, stable fixation, less operative trauma and early, active post-operative mobilization. The study compares two types of implant to determine efficacy in reduction and maintenance of reduction for fracture healing

ELIGIBILITY:
Inclusion Criteria:Patients who undergo hand surgery at University of Colorado Hospital and Denver Health Medical Center for surgical treatment of closed extraarticular metacarpal fracture(s). Fracture classification will be based off of AO Foundation/Orthopaedic Trauma Association guidelines and radiographic interpretation

* Non-operative Cohort: Patients who underwent non-operative management of closed extra-articular metacarpal fractures at both the University of Colorado and Denver Health Medical Center will also be reviewed.

Exclusion Criteria: Open metacarpal fractures (defined as any fracture associated with a laceration or break in skin continuity near the fracture site)

* Patients with previous history of metacarpal nonunion or malunion corrections on the affected digit
* Metacarpal fractures with intraarticular extension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo hand surgery at University of Colorado Hospital and Denver Health Medical Center for surgical treatment of closed extraarticular metacarpal fracture(s). Fracture classification will be based off of AO Foundation/Orthopaedic Trauma Association guidelines and radiographic interpretation
  • Non-operative Cohort: Patients who underwent non-operative management of closed extra-articular metacarpal fractures at both the University of Colorado and Denver Health Medical Center will also be reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Post-operative primary Outcomes | 30 Days
  Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) outcome measure score.

SECONDARY OUTCOMES:
Pain scale | 30-days
  Pain quantified on Graphic Rating Scale (GRS)
Measurement of range | 30-days
  Goniometer measurements of range of motion at metacarpophalangeal joint (MP), proximal interphalangeal joint (PIP), distal interphalangeal joint (DIP), in addition to any extensor lag at the MP joint.
Operative complications | 30-days
  Operative complications including but not limited to: bone nonunion and malunion, superficial and deep infections, hardware failure, stiffness, revision surgery and tendon adhesions/rupture.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Iorio, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol